CLINICAL TRIAL: NCT02339441
Title: Treatment Outcome in Early Diffuse Cutaneous Systemic Sclerosis
Acronym: ESOS
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof. Ariane herrick, Professor, University of Manchester
Other Study IDs: 10H101429
Record Dates: First submitted 2014-12-22; First posted 2015-01-15 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Early Diffuse Cutaneous Systemic Sclerosis
Keywords: Systemic sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Methotrexate; Mycophenolic Acid; Cyclophosphamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Methotrexate: Patients treated with Methotrexate at the entry of the study.
  Interventions: Drug: Methotrexate
- Mycophenolate Mofetil: Patients treated with Mycophenolate Mofetil at the entry of the study.
  Interventions: Drug: Mycophenolate mofetil
- Cyclophosphamide: Patients treated with Cyclophosphamide at the entry of the study
  Interventions: Drug: Cyclophosphamide
- No Immunosuppressant: Patients without immunosuppressant treatment at the entry of the study

INTERVENTIONS:
Drug: Methotrexate — Immunosuppressant agent. Patients treated with Methotrexate at the entry of the study, either oral or subcutaneous with a target dose of 20-25mg weekly.
  Groups: Methotrexate
Drug: Mycophenolate mofetil — Immunosuppressant agent. Patients treated with Methotrexate at the entry of the study,recommended dose 500 mg twice daily for 2 weeks increasing to 1gm twice daily.
  Groups: Mycophenolate Mofetil
Drug: Cyclophosphamide — Immunosuppressant agent. Patients treated with Methotrexate at the entry of the study, recommend use (i) IV. Minimum monthly dose 500mg/m2 with a recommended duration of 6-12 months. (ii) Oral. 1-2mg/day with a recommended duration of 12 months.
  Groups: Cyclophosphamide

SUMMARY:
The aim of the study is to compare the effectiveness of commonly used immunosuppressant treatments for early diffuse cutaneous systemic sclerosis (SSc).

DETAILED DESCRIPTION:
Diffuse cutaneous systemic sclerosis (SSc) is a rare autoimmune disease characterised by excessive connective tissue in the skin (causing skin thickening called 'scleroderma'), muscle, joints and internal organs. A number of different drugs with effects on the immune system (known as 'immunosuppressants') are currently being used by clinicians in the treatment of early diffuse cutaneous SSc, but all can have significant side effects. We want to know whether any one is definitely effective and, if so, which is the most effective.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 Skin thickening < 3 years Immunosuppressant use < 4 months Proximal skin involvement to face/neck, elbow or knee

Exclusion Criteria:

Previous use of more than 4 months of methotrexate, mycophenolate mofetil, cyclophosphamide or other immunosuppressive treatments

Previous use of immunosuppressant therapy other than methotrexate, mycophenolate mofetil or cyclophosphamide within previous months

Previous stem cell transplantation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibility:
  Age > 18 Skin thickening < 3 years Immunosuppressant use < 4 months Proximal skin involvement to face/neck, elbow or knee
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2010-06; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Skin score as measured by modified rodnan skin score | 24 months

SECONDARY OUTCOMES:
Pulmonary function as measured by right ventricular systolic pressure (RVSP) or pulmonary artery pressure (PAP) | 24 months
Echocardiographic findings | 24 months
Cochin hand function | 24 months
Fatigue as measured by the Functional Assessment of Chronic Illness Therapy (FACIT) scale | 24 months
Short form 36 questionnaire (SF-36) | 24 months
Scleroderma Health Assessment Questionnaire | 24 months
Haemoglobin | 24 months
Erythrocyte sedimentation rate | 24 months
Estimated glomerular filtration rate (eGFR) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Herrick, MD, phD, Principal Investigator — University of Manchester

REFERENCES:
- [Derived] Herrick AL, Peytrignet S, Lunt M, Pan X, Hesselstrand R, Mouthon L, Silman AJ, Dinsdale G, Brown E, Czirjak L, Distler JHW, Distler O, Fligelstone K, Gregory WJ, Ochiel R, Vonk MC, Ancuta C, Ong VH, Farge D, Hudson M, Matucci-Cerinic M, Balbir-Gurman A, Midtvedt O, Jobanputra P, Jordan AC, Stevens W, Moinzadeh P, Hall FC, Agard C, Anderson ME, Diot E, Madhok R, Akil M, Buch MH, Chung L, Damjanov NS, Gunawardena H, Lanyon P, Ahmad Y, Chakravarty K, Jacobsen S, MacGregor AJ, McHugh N, Muller-Ladner U, Riemekasten G, Becker M, Roddy J, Carreira PE, Fauchais AL, Hachulla E, Hamilton J, Inanc M, McLaren JS, van Laar JM, Pathare S, Proudman SM, Rudin A, Sahhar J, Coppere B, Serratrice C, Sheeran T, Veale DJ, Grange C, Trad GS, Denton CP. Patterns and predictors of skin score change in early diffuse systemic sclerosis from the European Scleroderma Observational Study. Ann Rheum Dis. 2018 Apr;77(4):563-570. doi: 10.1136/annrheumdis-2017-211912. Epub 2018 Jan 6. PMID 29306872
- [Derived] Herrick AL, Pan X, Peytrignet S, Lunt M, Hesselstrand R, Mouthon L, Silman A, Brown E, Czirjak L, Distler JHW, Distler O, Fligelstone K, Gregory WJ, Ochiel R, Vonk M, Ancuta C, Ong VH, Farge D, Hudson M, Matucci-Cerinic M, Balbir-Gurman A, Midtvedt O, Jordan AC, Jobanputra P, Stevens W, Moinzadeh P, Hall FC, Agard C, Anderson ME, Diot E, Madhok R, Akil M, Buch MH, Chung L, Damjanov N, Gunawardena H, Lanyon P, Ahmad Y, Chakravarty K, Jacobsen S, MacGregor AJ, McHugh N, Muller-Ladner U, Riemekasten G, Becker M, Roddy J, Carreira PE, Fauchais AL, Hachulla E, Hamilton J, Inanc M, McLaren JS, van Laar JM, Pathare S, Proudman S, Rudin A, Sahhar J, Coppere B, Serratrice C, Sheeran T, Veale DJ, Grange C, Trad GS, Denton CP. Treatment outcome in early diffuse cutaneous systemic sclerosis: the European Scleroderma Observational Study (ESOS). Ann Rheum Dis. 2017 Jul;76(7):1207-1218. doi: 10.1136/annrheumdis-2016-210503. Epub 2017 Feb 10. PMID 28188239